CLINICAL TRIAL: NCT02140008
Title: A Comparison of the I-gel and the Self-pressurised Air-Q Intubating Laryngeal Airway in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 1-2014-0011
Record Dates: First submitted 2014-05-12; First posted 2014-05-16 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: General Anesthesia; Supraglottic Airway Devices
Keywords: supraglottic airway devices; the i-gel; the self-pressurised air-Q intubating laryngeal airway,; children

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I-gel group (Experimental)
  Interventions: Device: Insertion of I-gel
- Air-Q group (Active Comparator)
  Interventions: Device: Insertion of air-Q

INTERVENTIONS:
Device: Insertion of I-gel — After induction of general anesthesia, I-gel will be inserted according to randomly allocated group.
  Arms: I-gel group
Device: Insertion of air-Q — After induction of general anesthesia, air-Q was inserted according to randomly allocated group.
  Arms: Air-Q group

SUMMARY:
Supraglottic airway devices (SADs) are well established in pediatric anesthetic practice. The pediatric i-gel and the self-pressurised air-Q (air-Q) are new supraglottic airway devices for children. The i-gel is made of a soft, gel-like elastomer with a noninflatable cuff. The air-Q is a new single-use device that may optimise the airway seal while reducing the potential for postoperative complications such as sore throat. The overall structure of the air-Q SP is identical to the original air-Q, except with regard to the inflatable cuff. The aim of this randomized trial was to compare the clinical performance of the i-gel and the air-Q SP.

ELIGIBILITY:
Inclusion Criteria:

* Children (1-108 month of age and 7-30kg) scheduled for elective surgery of short duration (less than 2 hr) undergoing general anesthesia using supraglottic airway

Exclusion Criteria:

* Patients with a potentially difficult airway, risk of aspiration such as gastroesophageal reflux disease, or active upper respiratory tract infection

Ages: 1 Month to 108 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2014-05; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
airway leak pressure | within 5 min after insertion of each device

SECONDARY OUTCOMES:
Insertion time (insertion parameter) | During and 1 min after insertion of each device
  insertion time was defined as the time from the attending anesthesiologist picking up the LMA until the confirmation on capnography.

OTHER OUTCOMES:
Ease of insertion (insertion parameter) | During and 1 min after insertion of each device
  Ease of insertion was graded from 1 to 4

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Seoul, Seoul, South Korea